CLINICAL TRIAL: NCT03573973
Title: Nudging Healthier Dietary Habits: Evaluation of a Supermarket Placement Strategy in the WRAPPED Study
Brief Title: Women's Responses to Adjusted Product Placement and Its Effects on Diet - 2
Acronym: WRAPPED2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Medical Research Council (Other Government); University of Southampton (Other); City, University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20986
Record Dates: First submitted 2018-04-25; First posted 2018-06-29 (Actual); Last update posted 2023-05-15 (Actual); Status verified 2022-05

CONDITIONS: Diet Modification
Keywords: Dietary inequalities; Public Health; Choice architecture; Supermarkets
MeSH Terms: interventions — Vegetables

STUDY DESIGN:
Intervention Model Description: Natural experiment with prospective matched controlled cluster design. The setting is a UK discount supermarket chain.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fresh fruit and vegetable placement intervention (Experimental): The intervention is a store refurbishment programme that includes the creation of a new fresh fruit and vegetable section at the store entrance with expanded range thus improving the availability and position of fresh fruit and vegetables.
  Interventions: Other: Improved product placement of fresh fruit and vegetables
- Control (Sham Comparator): The control condition is the existing store layout with a limited range of fresh fruit and vegetables that are placed at the back of the store.
  Interventions: Other: Sham comparator

INTERVENTIONS:
Other: Improved product placement of fresh fruit and vegetables — The intervention includes the creation of a new fresh fruit and vegetable section at the store entrance with expanded range thus improving the placement (availability and position) of fresh fruit and vegetables.
  Arms: Fresh fruit and vegetable placement intervention
Other: Sham comparator — The control condition is the existing store layout with a limited range of fresh fruit and vegetables that are placed at the back of the store.
  Arms: Control

SUMMARY:
This study is the largest supermarket trial internationally and will assess the effectiveness and cost-effectiveness of improving the placement of fresh fruit and vegetables in discount supermarkets in improving the fresh fruit and vegetable purchasing of women aged 18-45 years.

DETAILED DESCRIPTION:
WRAPPED2 (Women's Responses to Adjusted Product Placement and its Effects on Diet - 2) is a natural experiment with a prospective matched controlled cluster design. The setting is a discount supermarket chain in the United Kingdom regularly used by disadvantaged families for their main shop. The intervention is a store refurbishment programme that involves creation of a new fresh fruit and vegetable section in the store entrance. Control stores keep the existing layout with a limited range of fresh fruit and vegetables and placement of fresh fruit and vegetables at the back of the store.

A total of 45 participants will be recruited from each of 18 intervention and 18 matched control stores through the retailer's loyalty card scheme (postal letter) and shop floor recruitment; these methods proved effective during the pilot. Participants will be women aged 18-45 years who shopped at a study store in the 12 weeks before recruitment. This study is unique in its collection of individual level sales data, as well as demographic and dietary information, and is the first to collect outcome data for more than one family member. Participant's weekly sales data will be obtained through the retailer's loyalty card scheme and will cover 3 months before refurbishment, plus 0-3 months and 3-6 months after. Change in women's fresh fruit and vegetable purchasing from baseline to 3 months is the primary outcome. Secondary outcome data about women's diets, their young child's diet (2-6 years), food shopping habits, perceptions of supermarket environment, and psychosocial and demographic characteristics will be collected by telephone survey before refurbishment, and 1, 3 and 6 months after. Weekly sales data for study stores will be provided by the retailer.

Cost-effectiveness will be assessed from individual, retailer and societal perspectives. Process evaluation will assess implementation, mechanisms of impact and context.

This study is politically and scientifically important being one of the first field studies of this kind. The findings could provide strong evidence for future public health policy interventions to help address inequalities in diet and non-communicable disease risk by supporting development of a healthy store layout that could be adopted more widely in food retail outlets.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-60 years
* Hold a store loyalty card
* Shop regularly in a study store
* Shoppers who choose items in-store but opt for home delivery

Exclusion Criteria:

* Women under the age of 18 or over 60 years
* Males or children
* Irregular shopper or online-only shopper
* Do not hold store loyalty card

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 667 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Participant's weekly fruit and vegetable purchasing patterns | 0-6 month period post-refurbishment
  These data will be obtained through the retailer's loyalty card scheme and provide information about the number of items of each product purchased at each store visit.

SECONDARY OUTCOMES:
Women's dietary quality | 3 and 6 month follow-up post intervention commencement
  20-item food frequency questionnaire (FFQ) will be used to create standardised diet quality scores for each woman. A dietary quality score for each woman will be calculated by multiplying their reported frequency of consumption of each of the 20 items from their FFQ by corresponding weightings derived from the appropriate principal components analysis and then summing the results.
Children's dietary quality | 3 and 6 month follow-up post intervention commencement
  20-item food frequency questionnaire (FFQ) will be used to create standardised diet quality scores for each child. Dietary quality scores will be calculated by multiplying the reported frequency of consumption of each of the 20 items from their FFQ by corresponding weightings derived from the appropriate principal components analysis and then summing the results.
Women's daily fruit and vegetable intake | 3 and 6 months follow-up post intervention commencement
  2-item tool has been validated against urinary potassium and plasma ascorbic acid to describe high (≥5 portions/day) and low (≤2.5 portions/day) intake.
Weekly store sales of fresh fruit and vegetables | 0-3 and 0-6 month periods post-refurbishment
  Store sales data will be provided from electronic transaction records aggregated to the weekly level
To determine whether change in participants' in fruit and vegetable purchasing patterns (intervention effects) differ according to their level of educational attainment | 0-6 month period post-refurbishment
  To assess interaction on intervention effects according to participants' highest educational qualification attained in 3 groups (low=GCSE/school departure before 16 years of age, medium=A-levels/HND/diploma, high=degree)
Economic evaluation to assess the costs and benefits of the intervention from individual, retailer and societal perspectives | 6 month period post-refurbishment
  Use participant survey and purchasing data for food expenditure, time spent food shopping, as well as travel costs to and from supermarkets; retailer costs will be estimates generated through discussion with supermarket staff; societal costs will be estimated for resources associated with the capital investment, changes in food expenditure, time and travel costs for individuals and health and social care costs for diet-related health conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Univeristy of Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vogel C, Crozier S, Dhuria P, Shand C, Lawrence W, Cade J, Moon G, Lord J, Ball K, Cooper C, Baird J. Protocol of a natural experiment to evaluate a supermarket intervention to improve food purchasing and dietary behaviours of women (WRAPPED study) in England: a prospective matched controlled cluster design. BMJ Open. 2020 Feb 10;10(2):e036758. doi: 10.1136/bmjopen-2020-036758. PMID 32047023
- [Background] Muir S, Dhuria P, Roe E, Lawrence W, Baird J, Vogel C. UK government's new placement legislation is a 'good first step': a rapid qualitative analysis of consumer, business, enforcement and health stakeholder perspectives. BMC Med. 2023 Jan 26;21(1):33. doi: 10.1186/s12916-023-02726-9. PMID 36703194
- [Background] Muir S, Dhuria P, Vogel C. Government must proceed with landmark anti-obesity regulations in England. BMJ. 2022 Sep 30;378:o2358. doi: 10.1136/bmj.o2358. No abstract available. PMID 36180089
- [Derived] Baird J, Dhuria P, Payne H, Crozier S, Lawrence W, Vogel C. Implementation of a UK supermarket intervention to increase purchasing of fresh fruit and vegetables: process evaluation of the WRAPPED natural experiment. Int J Behav Nutr Phys Act. 2024 Nov 11;21(1):128. doi: 10.1186/s12966-024-01679-3. PMID 39529139